CLINICAL TRIAL: NCT04829838
Title: Comparison of Efficacy of Phenytoin With Levetireacetam for the Management of Children With Status Epilepticus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ayesha tariq (Other)
Collaborators: King Edward Medical University (Other)
Responsible Party: Sponsor-Investigator, ayesha tariq, Post graduate resident in Pediatrics medicine(MD Paeds), King Edward Medical University
Organization: King Edward Medical University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 700/RC/KEMU
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Status Epilepticus
Keywords: status epilepticus, children, phenytoin, levetireacetam
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous levetireacetam (Experimental): Drug:Intravenous levetireacetam will be given at a loading dose of 20-30mg/kg then it will be added in maintainance dose of (5-30mg/kg/day)
  Interventions: Drug: intravenous levetireacetam
- intravenous phenytoin (Experimental): Intravenous phenytoin will be given in loading dose of 20mg/kg then it will be added in maintainance dose i-e 5-8mg/kg/day
  Interventions: Drug: intravenous levetireacetam

INTERVENTIONS:
Drug: intravenous levetireacetam — phenytoin is considered as control drug in the study

SUMMARY:
The purpose of studyis to compare the efficacy of phenytoin with levetiracetam for the management of children with status epilepticus.Study performa consists of demographic variables,exclusion criteria,history of epilepsy and efficacy achieved or not.

DETAILED DESCRIPTION:
After getting informed consent 244 children with status epilepticus will be randomly classified into two groups.one group will receive levetireacetam and other group will be given phenytoin and their efficacy will be compared by observing them for breakthrough fits for next 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* childen of age less than 12 years either gender admitted in pediatric emergency with status epilepticus

Exclusion Criteria:

* children already taking either of trial drug or failed treatment with either of trial drug.children with comorbid conditions

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 244 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-07-26 (Estimated); Study Completion 2021-07-26 (Estimated)

PRIMARY OUTCOMES:
comparison of efficacy of levetireacetam with phenytoin for the management of children with status epilepticus | 48 hours
  the intervention will be considered efficacious if child will not have breakthrough fits for 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Haroon Hamid, MBBS,FCPS, Principal Investigator — King Edward Medical University
Locations (1):
- Ayesha Tariq, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Smith DM, McGinnis EL, Walleigh DJ, Abend NS. Management of Status Epilepticus in Children. J Clin Med. 2016 Apr 13;5(4):47. doi: 10.3390/jcm5040047. PMID 27089373
- [Background] Abend NS, Loddenkemper T. Pediatric status epilepticus management. Curr Opin Pediatr. 2014 Dec;26(6):668-74. doi: 10.1097/MOP.0000000000000154. PMID 25304961